CLINICAL TRIAL: NCT03735433
Title: The Effect of 81mg vs 162mg ASA for Preeclampsia Prevention in Obese Women at High Risk for Developing Preeclampsia
Brief Title: The Effect of Two Aspirin Dosing Strategies for Obese Women at High Risk for Preeclampsia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: futility
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kara M Rood, MD, Prinicple Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBASA
Record Dates: First submitted 2018-11-04; First posted 2018-11-08 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Preeclampsia
Keywords: aspirin; obesity
MeSH Terms: conditions — Pre-Eclampsia; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 81 mg daily aspirin dose (No Intervention): obese women >30 BMI at risk for preeclampsia will receive recommended 81mg ASA
- 162mg daily aspirin dose (Active Comparator): obese women >30 BMI at risk for preeclampsia will receive increased dose of 162mg ASA
  Interventions: Drug: 162mg aspirin dose

INTERVENTIONS:
Drug: 162mg aspirin dose — 2 pills of 81mg aspirin
  Arms: 162mg daily aspirin dose

SUMMARY:
Low dose aspirin (LDA) is used for preeclampsia (PE) prevention in high risk women, but the precise mechanism and optimal dose is not known. Evidence in the non-obstetric literature suggests AR may be more common among patients with a high body mass index (BMI). Recent unpublished data showed that LDA substantially lowers TxB2 levels regardless of BMI, but rates of complete platelet inhibition are lower in women with BMI ≥40. This data suggests that higher doses of ASA may be necessary in obese women. Therefore we plan determine if use of 162mg compared to the traditional 81mg ASA decreased rates of preeclampsia in women considered high risk for developing preclampsia.

DETAILED DESCRIPTION:
Evidence suggests that an imbalance in prostacyclin and thromboxane A2 (TxA2) plays a key role in PE. Aspirin (ASA) has a dose-dependent effect blocking production of TxA2, a potent stimulator of platelet aggregation (PA) and promoter of vasoconstriction. Incomplete inhibition of PA, designated aspirin resistance (AR), can be reduced by increasing the ASA dose.

ELIGIBILITY:
Inclusion Criteria:

* BMI at enrollment >/= 30
* plan for ASA for preeclampsia prevention

Exclusion Criteria:

* BMI < 30
* already on ASA

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 152 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State Medical Center Labor and Delivery Unit, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 81 mg Daily Aspirin Dose | 162mg Daily Aspirin Dose
Started | 76 | 76
Completed | 0 | 0
Not Completed | 76 | 76

BASELINE CHARACTERISTICS:
Population: Baseline analysis population data was not obtained as we did not complete this study. No baseline data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | 81 mg Daily Aspirin Dose | 162mg Daily Aspirin Dose | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Diagnosis of Preeclampsia
Description: by acog definitions
Time Frame: Through study completion, an average for 10 months
Population: Study outcomes were not collected as no participants completed either 81 mg or 162 mg aspirin dose. Participation was terminated before completion of the study.
Arm/Group | 81 mg Daily Aspirin Dose | 162mg Daily Aspirin Dose
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Aspirin Resistance Based on Incomplete Inhibition of TBx2
Description: incomplete platelet inhibition measured by urinary TBx2
Time Frame: Through study completion, an average for 10 months
Population: as for outcome 1
Arm/Group | 81 mg Daily Aspirin Dose | 162mg Daily Aspirin Dose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average for 10 months
Arm/Group | 81 mg Daily Aspirin Dose | 162mg Daily Aspirin Dose
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/76 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT03735433/Prot_SAP_000.pdf